CLINICAL TRIAL: NCT06992791
Title: Labor Education to Reduce Postpartum Traumatic Stress: A Randomized Controlled Trial
Brief Title: Labor Education to Reduce Postpartum Traumatic Stress
Acronym: LEPT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Nicole Teal, Assistant Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 812358
Record Dates: First submitted 2025-04-30; First posted 2025-05-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Complication; Posttraumatic Stress Symptoms
Keywords: Posttraumatic stress disorder; Childbirth related PTSD; prenatal education; traumatic childbirth; Posttraumatic stress syndrome
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prenatal Education Arm (Experimental): Those in Group 1 (intervention group) will be given access to intrapartum education videos provided by Tinyhood between 30weeks and delivery.
  Interventions: Behavioral: Prenatal Education on Childbirth
- Control Arm (No Intervention): Those in the control arm will be given a series of surveys administered by RedCap, and will continue with standard prenatal care. These participants will also have access to community prenatal education classes.

INTERVENTIONS:
Behavioral: Prenatal Education on Childbirth — Starting at 30 weeks, participants will be given access to Tinyhood, an online educational service aimed at perinatal education. Text reminders will be sent periodically throughout the third trimester to encourage interaction with educational videos and written materials, which will be tracked for number of interactions via the Tinyhyood interface. The videos include: "Pregnancy Milestones", "Physically and Mentally Preparing for Labor", "Finding Support During Labor", "Deciding Birth Preferences and Self-Advocacy", "Signs Labor Is Approaching", "Contractions", "Signs of Preterm Labor", "Going to the Hospital", "Baby's Positioning", "Stages of Labor", "Induction of Labor", "Managing Pain", "Pain Options in Labor", "Relaxation Techniques for Labor", " Breathing Techniques", "Labor Positions" and several handouts highlighting common obstetrical emergencies and possible interventions.
  Arms: Prenatal Education Arm

SUMMARY:
The goal of this randomized controlled trial is determine if education on common events in labor in nulliparous women can reduce the postpartum traumatic symptoms. The main question it aims to answer are:

* Does prenatal education on labor events reduce post-traumatic symptoms, as measured by thePost Traumatic Stress Disorder Cecklist for Diagnostic and Statistical Manual for Mental Health Disorders (PCL-5) at 6 weeks postpartum?
* Does prenatal education on labor affect labor outcomes?

Participants will be given surveys:

* At enrollment on mental health and previous traumatic experiences
* After education on expectations on childbirth
* After delivery on experience of childbirth
* At 6 weeks and 6 months postpartum on traumatic symptoms and mental health outcomes.

They will also have the option to participate in collection of discarded cerebrospinal fluid, blood and serum and physiologic sensitivity testing.

DETAILED DESCRIPTION:
Hypothesis:

This randomized trial was designed to determine if prenatal education on intrapartum experiences reduces postpartum trauma symptoms compared to standard prenatal care.

Methods and Procedures:

1. Identification. Participants will be identified by reviewing prenatal care providers (midwives, generalist obstetricians and perinatology) schedules for those that meet the inclusion criteria and approached in person at ultrasound or clinic appointments to be offered participation. Consent will be obtained at this time. Patient may also be called between appointments, and consent will be signed via HIPAA compliant REDCap.
2. Randomization. Participants will be randomized 1:1 to one of the two study groups described below. Neither participants or medical providers will be blinded to the randomization group. The randomization will be done using the block randomization module in REDcap.
3. Intervention: For those in Group 1, starting at 30 weeks they will be contacted by email and text to provide links to online education videos on intrapartum experiences. Patients will receive text reminders in the third trimester to encourage interaction with the videos, and interaction will be tracked online.
4. Collection of health information. The medical record of the pregnant person and the neonate will be used to collect information related to the pregnancy, delivery, and immediate post-delivery care into REDCap database. Baseline characteristics will include demographic information, prenatal care details such as type of provider, gestational age which established care, visit types, maternal medical conditions and obstetric history. Delivery characteristics will include labor characteristics (length of labor, gestational age, fetal heart rate tracings, any interventions in labor, mode of delivery and newborn and maternal complications during delivery admission).
5. Survey Administration. All participant will be give the same surveys on the same time scales. At enrollment, participants will be given a series of surveys on baseline mental health outcomes (Primary Care PTSD for DSM-5, Generalized Anxiety Disorder -7, Edinburgh Postnatal Depression Scale, Adverse Childhood Experiences), social experiences (Everyday Discrimination scale) and expectations for childbirth (Wijma Delivery Expectations Questionnaire (W-DEQ) on a iPad in clinic. Participants will be contacted via text and/or email for a repeat W-DEQ scale at term and after delivery. They will be contacted again via text and/or email at six weeks postpartum with 2 reminders if not replied (survey open 6 weeks-12 weeks) postpartum, and then again six months (with two reminders, survey open to 8 months) postpartum. All of these surveys will be administered by RedCap and collected securely.
6. Collection of specimens. Cerebrospinal fluid will only be collected from patients who are already undergoing dural puncture as standard of care for their anesthesia plan. Usual standard of care for epidural anesthesia at our hospital is to perform a dural puncture at the time of epidural placement which results in 0.5-1 mL of cerebrospinal fluid release through the needle used to place the epidural. Instead of allowing this fluid to be discarded, we will collect it in sterile tubes. The anesthesia plan will in no way be impacted by our study. If the anesthesia team at the time of placement feels a dural puncture is not appropriate, then the dural space will not be entered and fluid will not be collected. The sample collected will not exceed the amount that would be discarded as waste in a routine procedure and will be collected in a sterile fashion, presenting no additional risk to patients. Additionally, up to 1 cc discarded urine from foley catheter drainage, and up to 1 cc of additional blood will be taken at the time of already scheduled blood draws. No additional blood draws or urine samples will be requested outside of routine care. Stool collection kits will also be given to participants on L&D to collect if able, with instructions on how to collect stool off toilet paper and return samples. This will be used to create a biospecimen repository with no genetic or identifying information.
7. Physiologic testing. A subgroup of participants will undergo cutaneous mechanical sensitivity assays, radiant heat assays and pressure sensitivity assays. The cutaneous mechanical sensitivity testing involves stimulation with von Frey filaments to determine the size of filament that the participant can detect. The heat sensitivity assay will be preformed a radiant heat devices that uses a focused light beam to slowly heat a participants skin through safety glass, with participants indicating first when temperature is detected and in a second trial, when it becomes painful. This was assembled according to the protocol attached, using the IITC Plantar Analgesia Meter assembled in the attached protocol using a Hargraves testing platform. The heat assay assessing constant temperature will apply a stimulus for 3 seconds and request rating of pain, set at the typical minimal stimulus required to feel pain. The pressure sensitivity assay involves a 2 cm probe pressed against participant skin until they identify the threshold where it becomes painful. The probe is a standard clinical threshold algometer, as shown in the picture. For all of these assays, they will be tested on the right and left forearm, and right and left calf. These will be done at admission to labor and delivery, and patients have can opt out without impacting survey collection. A convenience sample will be collected when researchers are available on labor and delivery (typically 10 am to 6 pm), expecting to be no more than 20% of the enrolled population to be captured at delivery admission. Patients will be approached if they are early in their admission, have not yet requested an epidural and have not opt-ed out to either biospecimen collection or physiologic testing.

ELIGIBILITY:
Inclusion criteria:

* Maternal age > 18 years
* Nulliparous
* Singleton pregnancy between 18-30 weeks
* English Speaking

Exclusion criteria:

* Prenatal care outside of UCSD
* Plan to deliver outside of UCSD
* Contraindications to vaginal delivery at time of enrollment
* Major fetal anomalies at time of Level II Ultrasound
* No access to smart phone and/or internet

Ages: 18 Years to 51 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-10-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Post-traumatic stress disorder checklist for Diagnostic and Statistical Manual of Mental Health Disorders-5 (PCL-5) | 6-12 weeks postpartum
  Validated measurement for PTSD, scores 0-80 with higher being more symptomatic

SECONDARY OUTCOMES:
Change in Fear of Childbirth as measured by Wijma Delivery Experience Form A | At enrollment and at 36-38 weeks of pregnancy
  A change in scores over the third trimester using wijma Delivery Expectations Form A, a validated scale on expectations and delivery experiences with scores from 0-165, with higher scores indicating more fear of childbirth
Post-traumatic stress disorder checklist for Diagnostic Statistics and Mental Health Manual-5 (PCL 5) | 6-8 months postpartum
  Validated measure of PTSD assessment, scores 0-80 with higher being more symptomatic over a longer time frame
Delivery Experience as measured by Wijma Delivery Experience Form B | 0-2 weeks postpartum
  Wijma Delivery Expectations Form B, a validated scale on expectations and delivery experiences with scores from 0-165, with higher scores indicating more fear of childbirth
Rate of Labor Interventions | At delivery
  Chart review recording the rate of labor interventions, including amniotomy, induction, epidural, doula use, and pitocin at delivery admission
Rate of Obstetric Complications | 0-6 weeks after delivery admission
  Chart review recording the rate of composite of adverse obstetric outcomes including postpartum hemorrhage, shoulder dystocia, cesarean delivery or operative delivery and indication, development of venous thromboembolism, obstetric anal sphincter injuries, hysterectomy, intensive care unit admission or death
Postpartum Depression as assessed by Edinburgh Postnatal Depression Screen | 6 weeks - 12 weeks postpartum
  EPDS (Edinburg Postnatal Depression Screen) is a validated survey for pre and postnatal depression, with scores ranging from 0-30 with higher score indicating increased symptom burden
Postpartum Depression as assessed by Edinburgh Postnatal Depression Screen | 6 months to 8 months postpartum
  EPDS (Edinburg Postnatal Depression Screen) is a validated survey for pre and postnatal depression, with scores ranging from 0-30 with higher score indicating increased symptom burden with a second outcome at a longer time scale
Postpartum Anxiety as assessed by Generalized Anxiety Disorder - 7 item (GAD-7) | 6 weeks - 12 weeks postpartum
  GAD-7 is a validated survey for anxiety, with scores ranging from 0-21 with higher score indicating increased symptom burden
Postpartum Anxiety as assessed by Generalized Anxiety Disorder - 7 item (GAD-7) | 6 months to 8 months postpartum
  GAD-7 is a validated survey for anxiety, with scores ranging from 0-21 with higher score indicating increased symptom burden

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact rwiley@health.ucsd.edu
URL: https://blink.ucsd.edu/research/policies-compliance-ethics/compliance/research_data_policy.html

REFERENCES:
- [Background] Kostek M, Polaski A, Kolber B, Ramsey A, Kranjec A, Szucs K. A Protocol of Manual Tests to Measure Sensation and Pain in Humans. J Vis Exp. 2016 Dec 19;(118):54130. doi: 10.3791/54130. PMID 28060280
- [Background] Horsch A, Garthus-Niegel S, Ayers S, Chandra P, Hartmann K, Vaisbuch E, Lalor J. Childbirth-related posttraumatic stress disorder: definition, risk factors, pathophysiology, diagnosis, prevention, and treatment. Am J Obstet Gynecol. 2024 Mar;230(3S):S1116-S1127. doi: 10.1016/j.ajog.2023.09.089. Epub 2024 Jan 9. PMID 38233316